CLINICAL TRIAL: NCT02973906
Title: Comparing Web, Group, and Telehealth Formats of a Military Parenting Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1407S52001
Record Dates: First submitted 2015-05-04; First posted 2016-11-28 (Estimated); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Parenting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ADAPT Self Directed web (Other): ADAPT Self Directed Web. In the self-directed web-only ADAPT condition, participants have access to the full ADAPT website (10 modules, online discussion forum)
  Interventions: Other: ADAPT Self Directed web
- ADAPT individualized web-facilitated (Other): This condition comprises access to the full ADAPT web program with augmentation of individual facilitator web support (i.e. the facilitator connects via Google Hangout). Facilitators meet with families at a mutually convenient time weekly (10-14 weeks, approximately 3 sessions per month).
  Interventions: Other: ADAPT individualized web-facilitated
- Group-based ADAPT (Other): Groups will meet weekly for 120 minutes, at a time convenient to participants (usually early evening). Groups cover core ADAPT/PMTO topics
  Interventions: Other: Group-based ADAPT

INTERVENTIONS:
Other: ADAPT Self Directed web — In the self-directed web-only ADAPT condition, participants have access to the full ADAPT website (10 modules, online discussion forum
  Arms: ADAPT Self Directed web
Other: ADAPT individualized web-facilitated — This condition comprises access to the full ADAPT web program as described above, with augmentation of individual facilitator web support (i.e. the facilitator connects via Google Hangout). Facilitators meet with families at a mutually convenient time weekly (10-14 weeks, approximately 3 sessions per month).
  Arms: ADAPT individualized web-facilitated
Other: Group-based ADAPT — Groups will meet weekly for 120 minutes, at a time convenient to participants (usually early evening). Groups cover core ADAPT/PMTO topics:
  Arms: Group-based ADAPT

SUMMARY:
The overarching goal of this study is to advance research on family-based prevention of negative child outcomes for reintegrating Operation Enduring Freedom/Operation Iraqi Freedom personnel by evaluating different formats of a parenting program, After Deployment, Adaptive Parenting Tools (ADAPT). The ADAPT program is based upon the Parent Management Training-Oregon Model/PMTO, but adapted for military deployed families. The PI will examine which of three delivery formats of ADAPT is most effective at reducing youth risk behaviors associated with negative childhood outcomes by improving parenting, child, and parent adjustment. There is a clear intent to benefit all subjects in this study (except surveyed teachers), including children.

DETAILED DESCRIPTION:
The overarching goal of this study is to advance research on family-based prevention of negative child outcomes for reintegrating Operation Enduring Freedom/Operation Iraqi Freedom personnel by evaluating different formats of a parenting program, After Deployment, Adaptive Parenting Tools (ADAPT). The ADAPT program is based upon the Parent Management Training-Oregon Model/PMTO, but adapted for military deployed families. The investigators will examine which of three delivery formats of ADAPT is most effective at reducing youth risk behaviors associated with negative childhood outcomes by improving parenting, child, and parent adjustment. There is a clear intent to benefit all subjects in this study (except surveyed teachers), including children.

Combat deployment and related challenges are family stressors, associated with more negative parent-child interactions, ineffective and coercive parenting practices and lower levels of parenting satisfaction. Disrupted parenting practices are well-known predictors of risk for child adjustment difficulties that are precursors to youth substance use, including behavior problems, school failure, deviant peer association, and depression . These child adjustment problems can contribute to continuing parental stress, increasing parental distress, and further disrupting parenting.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria are:

* one parent has returned from deployment to OIF or OEF
* at least one child ages 5-12 in their custody and living with parent(s) in the home
* high speed internet access at home We will include both single-and two-parent families, as well as families where care is shared between non-partnered adults (e.g. grandparent and mother)

Exclusion Criteria:

* active psychosis
* an open child protection case for abuse or neglect in the family
* a serious child mental health diagnosis
* families who piloted material or participated in or are currently participating in the original ADAPT RCT.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Change in parenting practices and parent/child interactions | Change from Baseline, 6 months, 12 months, 24 months
  Observed parenting is coded using FIT (Family Interaction Task) and self-report of parenting using the APQ (Alabama parenting Questionnaire),

SECONDARY OUTCOMES:
Change in child adjustment and substance use | Change from Baseline, 6 months, 12 months, 24 months
  Child adjustment assessed using BASC-2 (teacher, parent, and child self-report); Child intentions and use of substances assess using the Alcohol Use Intentions and Behavior Scale; Child distress measured by CDI (Children's Depression Inventory); Child peer adjustment is measured by 16-item scale assessing loneliness and dissatisfaction with peer relations; Deviant peer association measured using "Describing Friends"
Change in parenting stress and support | Change from Baseline, 6 months, 12 months, 24 months
  Parenting Stress Index-Short Form
Participant report of satisfaction with intervention | Change from Baseline, 6 months, 12 months, 24 months
  Two 10-item measures: (1) group satisfaction and (2) online satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Gweitrz, PhD, Principal Investigator — Institute for Translational Research in Children's Mental Health University of Minnesota
Locations (1):
- Institute for Translational Research in Children's Mental Health, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2018-05-04): https://cdn.clinicaltrials.gov/large-docs/06/NCT02973906/Prot_001.pdf